CLINICAL TRIAL: NCT01539109
Title: Improving Spinal Cord Injury Rehabilitation Interventions by Retraining the Brain With Stimulation: Applying Concepts From Stroke
Brief Title: Improving Spinal Cord Injury Rehabilitation Interventions by Retraining the Brain With Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Telemedicine & Advanced Technology Research Center (Other)
Responsible Party: Principal Investigator, Ela B. Plow, Project Scientist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-334; RPC 2016-195 (Other Grant/Funding Number: Conquer Paralysis Now)
Record Dates: First submitted 2012-02-16; First posted 2012-02-27 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Spinal Cord Injury
Keywords: Incomplete Spinal Cord Injury; Quadriplegia; Tetraplegia; SCI; Spinal Cord Disease; Spinal Cord Injury; iSCI; Transcranial Direct Current Stimulation; tDCS; SCI recovery; brain stimulation; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Spinal Cord Diseases | interventions — Rehabilitation; Transcranial Direct Current Stimulation; Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehab and tDCS (Experimental): Patients in this group will receive Noninvasive brain stimulation: tDCS, during rehabilitation exercises of the weak upper limbs for 2 hours per day, 5 times a week, for 2 weeks. tDCS is Transcranial Direct Current Stimulation. Prior to this 2-week intervention phase, all patients will be monitored over a 2-week control phase.
  Interventions: Behavioral: Rehabilitation; Procedure: Noninvasive brain stimulation: tDCS
- Rehab and sham tDCS (Sham Comparator): Patients in this group will receive Sham tDCS: placebo noninvasive brain stimulation, during rehabilitation exercises of the weak upper limbs for 2 hours per day, 5 times a week, for 2 weeks. tDCS is Transcranial Direct Current Stimulation. Prior to this 2-week intervention phase, all patients will be monitored over a 2-week control phase
  Interventions: Behavioral: Rehabilitation; Procedure: Sham tDCS: placebo noninvasive brain stimulation

INTERVENTIONS:
Behavioral: Rehabilitation — Patients will receive training upon tasks of daily living. Patients will perform these exercises in our laboratory under the supervision of qualified personnel.
Procedure: Noninvasive brain stimulation: tDCS — TDCS is a method of noninvasive stimulation of the brain. Using electrodes placed in saline-soaked sponges, low level of direct current (2mA) is delivered over the scalp. This intervention is considered safe and noninvasive because it does not involve implantation or injection or any skin penetration. In the present study, tDCS will be delivered to patients in the experimental group for 2 hr each day for 5 days a week for 2 weeks in conjunction with therapy for the affected hand.
  Other Names: tDCS; Transcranial Stimulation; Transcranial Direct Current Stimulation; Brain stimulation
  Arms: Rehab and tDCS
Procedure: Sham tDCS: placebo noninvasive brain stimulation — Placebo set-up for noninvasive brain stimulation will be similar to that for the active tDCS; sponge electrodes would be placed on the scalp and connected to a batter-operated device. Patients will not receive the effective level of direct current as would delivered in active tDCS intervention. But patients will not be able to decipher whether they are receiving active or placebo tDCS.
  Other Names: sham tDCS; placebo tDCS
  Arms: Rehab and sham tDCS

SUMMARY:
The purpose of this study is to investigate whether combining a noninvasive method of brain stimulation, called Transcranial Direct Current Stimulation (tDCS), enhances the effect of training of the affected upper limbs in patients with incomplete Spinal Cord Injury.

DETAILED DESCRIPTION:
The long-term objective of this study is to optimize the rehabilitative potential in spinal cord injury (SCI) by maximally harnessing the potential available for functional neural plasticity. SCI is an important cause of serious, long-term disability in young adults. This fact, further complicated by rising disability-related costs, makes SCI a significant economic and social burden. Upper limb dysfunction is one of the most prevalent and debilitating impairments. More than 75% of patients with quadriplegia (paralysis of all 4 limbs following spinal cord injury in neck and upper back) prioritize return of upper limb function over any other lost function. Alleviating deficits of the upper limb may represent a cost-effective stategy to reducing the burden of SCI.

Although various exercise programs and neuromuscular stimulation methods have been employed to mitigate functional impairments of the arm and hand, success of these modalities is still debated. Evidence for efficacy of rehabilitation is inconclusive as outcomes are variable, confounded by methodological issues, and have shown poor generalizability. It is now speculated that limited succcess of rehabilitation emerges from inability of current methods to adequately harness the potential for significant neuroplasticity available in SCI.

Even though the site of damage in SCI does not involve the brain, the neural networks in the brain that control movement of the arm and hand are markedly affected. These regions lose their territory that the investigators argue could hamper effects of upper limb therapy. The Investigators objective is to directly modulate adaptive plasticity in these regions of the brain to enhance function of the upper limb in iSCI. The Investigators central hypothesis is that noninvasive brain stimulation, called transcranial direct current stimulation (tDCS), when delivered concurrently with rehabilitation will generate synergistic functional advantage. Adaptive plasticty would be obeserved as changes in structure of pathways emerging from the brain and the individual's function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with incomplete spinal cord injury (iSCI) that occurred at least 6 months ago

Exclusion Criteria:

* History of epilepsy in a first degree relative
* Use of anticonvulsants
* Pregnant
* Implanted pumps, shunts, or neurostimulators
* Neurologic condition affecting sensorimotor systems
* Brain tumor
* Dementia
* Substance abuse
* Stroke
* Damaged skin on the scalp
* Concurrent upper limb rehabilitation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in Upper Limb Function from Baseline | Strength, activities and impairments will be measured at The patient will receive TMS during at baseline, post-2 weeks, post-4 weeks and 3-month followup
  Upper limb function will be measured by the Upper Extremity Motor Score (UEMS), capacity tasks in the form of the Grasp and Release Task (GRT) test, and pinch grip impariment that will be measured by a maximum voluntary isometric pinch force.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) of the brain | The patient will receive MRI during at baseline, post-2 weeks, and post-4 weeks
  MRI will be used to measure changes in structure of the brain and its pathways as a result of training
Physiology of Brain studied with Noninvasive Brain Stimulation using Transcranial Magnetic Stimulation (TMS) | The patient will receive TMS during at baseline, post-2 weeks, and post-4 weeks
  TMS is a noninvasive technique of brain stimulation that examines the activity of regions of brain devoted to movement. Without implanting, or injecting or penetrating the brain, simply by using scalp-based recordings, TMS can assess functionality of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Ela B Plow, PhD PT, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The Investigator not be sharing or releasing any study data to third parties outside the Cleveland Clinic

REFERENCES:
- [Derived] Potter-Baker KA, Janini DP, Lin YL, Sankarasubramanian V, Cunningham DA, Varnerin NM, Chabra P, Kilgore KL, Richmond MA, Frost FS, Plow EB. Transcranial direct current stimulation (tDCS) paired with massed practice training to promote adaptive plasticity and motor recovery in chronic incomplete tetraplegia: A pilot study. J Spinal Cord Med. 2018 Sep;41(5):503-517. doi: 10.1080/10790268.2017.1361562. Epub 2017 Aug 7. PMID 28784042